CLINICAL TRIAL: NCT07257614
Title: Left Atrial Appendage Occlusion in Dialysis Patients With Atrial Fibrillation: A Multicentre Pilot Study
Acronym: LAAO-DAF
Status: Not yet recruiting | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: The Queen Elizabeth Hospital (Other); Pok Oi Hospital (Other); Tuen Mun Hospital (Other Government); Princess Margaret Hospital, Hong Kong (Other Government); Alice Ho Miu Ling Nethersole Hospital (Other); Kiang Wu Hospital (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical Assistant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2025.630
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Dialysis; Chronic Kidney Disease (Stages 3b-5); Atrial Fibrillation; End Stage Kidney Failure; Stroke Prevention in Patients With Atrial Fibrillation; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Renal Insufficiency, Chronic; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Eligible participants, aged ≥18 with documented AF and ESRF on peritoneal dialysis (PD) or hemodialysis (HD), will undergo LAAO using the Watchman Flx PRO device, follow-up for 1 year post-operation to track their outcome
- Retrospective cohort: Comparison of clinical outcomes (1 year stroke/TIA, major bleeding and CV death) with matched cohort identified from exisiting dialysis registry will be conducted.

SUMMARY:
Objectives: This pilot study aims to evaluate the safety and efficacy of left atrial appendage occlusion (LAAO) in dialysis patients and atrial fibrillation (AF) to establish a novel stroke prevention strategy and determine an optimal post-occlusion antithrombotic regime. Page 3 of 50 Hypothesis: The study tests the hypotheses that LAAO is safe for dialysis patients, that a single antiplatelet regimen postprocedure is safe, and that LAAO effectively reduces the composite endpoint of stroke/transient ischemic attack and major bleeding compared to standard care. Instruments: The study employs a multicenter, single-arm prospective registry design. Eligible participants, aged ≥18 with documented AF and ESRF on peritoneal dialysis (PD) or hemodialysis (HD), will undergo LAAO using the Watchman Flx PRO device. Propensity score matched historical cohort from dialysis registry will be identified for comparison.

Main Outcome Measures: The primary endpoint is the composite of stroke/transient ischemic attack/systemic embolism and non-procedural-related major bleeding at one year. Secondary endpoints include individual rates of these events, procedural safety and device occlusion effectiveness. Data Analysis and Expected Results: Statistical analysis will involve descriptive statistics, chi-squared tests, and propensity score matching. A p-value of <0.05 will be deemed significant. The pilot study anticipates a low peri-procedural complication rate (≤5%) and confirms LAAO's efficacy in stroke and major bleeding reduction in Chinese PD and HD patients compared to standard care. This data will inform the design of a larger randomized controlled trial aimed at validating LAAO as a safe alternative for AF management in dialysis populations.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* End stage renal failure on peritoneal dialysis or haemodialysis
* documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation;
* CHADS2-VASc >=2
* The patient is willing and able to comply with the required medication post-procedure and follow-up evaluations;
* Able to consent

Exclusion Criteria:

* Patients who require long-term anticoagulation for a condition other than AF, e.g. pulmonary embolism, deep vein thrombosis, anti-phospholipid syndrome
* Mechanical valve replacement
* Active infection with bacteraemia;
* Pregnant or nursing patients and those who plan pregnancy during the study period. Female patients of childbearing potential must have a negative pregnancy
* Known hypersensitivity or contraindication to aspirin, clopidogrel, heparin, any device material or component (nickel titanium, PET, polypropylene), and/or contrast;
* Left atrial appendage is obliterated and surgical ligated;
* Underwent any cardiac or non-cardiac interventional or surgical procedure within 30 days prior to the procedure or planned to have the interventional or surgical procedure within 60 days after implant procedure (e.g., cardioversion, ablation, percutaneous coronary intervention, etc.);
* Recent (within 90 days prior to procedure) stroke, transient ischemic attack, or myocardial infarction;
* New York Heart Association Class IV;
* Life expectancy is less than 1 year;
* Current participation in another investigational drug or device study.
* Echocardiogram exclusion:

  i. Moderate mitral stenosis or above ii. LVEF <30% iii. Intracardiac thrombus iv. Presence of a cardiac tumour. v. Existing circumferential pericardial effusion >5 mm; vi. Presence of a high-risk Patent Foramen Ovale (PFO), defined as an atrial septal aneurysm (excursion >15 mm or length >15 mm) or large shunt (early, within 3 beats and/or substantial passage of 20 bubbles)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study employs a multicenter, single-arm prospective registry design. Eligible participants, aged ≥18 with documented AF and ESRF on peritoneal dialysis (PD) or hemodialysis (HD), will undergo LAAO using the Watchman Flx PRO device. Propensity score matched historical cohort from dialysis registry will be identified for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
1 year transient ischemic attack | 1 year
  Rate of transient ischemic attack in enrolled patient at 1 year
1 year stroke rate | 1 year
  Stroke rate of enrolled cases at 1-yera follow-up
1 year major bleeding rate | 1 year
  Rate of major bleeding (BRAC 3-5) of enrolled cases at 1-year follow-up

SECONDARY OUTCOMES:
1 year systemic embolism rate | 1 year
  Rate of systemic embolism in enrolled patient at 1 year
1 year minor bleeding rate | 1 year
  Rate of minor bleeding (BRAC 1-2) in enrolled patient at 1 year
LAAO safety endpoint | 7 days post-discharge
  occurrence of death between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of ischemic stroke between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of systemic embolism between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of device-related events requiring open cardiac surgery between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of device-related events requiring major endovascular intervention between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of procedure-related events requiring open cardiac surgery between the time of implant and within 7 days after hospital discharge
LAAO safety endpoint | 7 days post-discharge
  occurrence of procedure-related events requiring major endovascular intervention between the time of implant and within 7 days after hospital discharge
LAAO effectiveness endpoint | 1 year
  The incidence of effective LAA closure, defined as any peri-device flow ≤5 mm per core laboratory-assessed CT at 1 year
Peri-device leak rate at 1 month | 1 month
  Major Peri-Device Leak (>5mm) at 1 month follow-upr
Device Related Thrombus rate at 1 month | 1 month
  Device Related Thrombus at 1 month follow-up
Rate of device endotheliasation at 1 month | 1 month
  Rate of device endotheliasation at 1 month follow-up CT
Rate of device endotheliasation at 3 month | 3 month
  Rate of device endotheliasation at 3 month follow-up CT
Rate of device endotheliasation at 12 month | 12 month
  Rate of device endotheliasation at 12 month follow-up CT
Rate of 1-year cardiovascular mortality at 12 month | 12 month
  Rate of 1-year cardiovascular mortality in enrolled cases at 12 month follow-up
Comparison of outcome between prospective and retrospective group | 12 month
  Comparison of clinical outcome with matched cohort identified from dialysis registry will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Chak Yu So, Clinical Assistant Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese Universityy of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No